CLINICAL TRIAL: NCT05089825
Title: Cervical Cancer Screening: Evaluation of Telehealth to Enhance HPV Self-Collection
Brief Title: Telehealth & HPV Self-Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Amanda Bruegl, MD, Clinical Instructor, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00023478; OHSU IRB 23478 (Other: OHSU Institutional Review Board)
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Gynecologic Cancer
Keywords: Pap Smear; Human papillomavirus; Telehealth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receive routine instructions (Active Comparator): Participants will receive routine instructions included in the myLAB Box Clinical Laboratory Improvement Amendments (CLIA) certified collection kit
  Interventions: Other: Receive routine instructions
- Telehealth Visit (Active Comparator): Participants will have a telehealth-based instructional visit and receive routine instructions included in the myLAB Box commercially available, CLIA certified collection kit
  Interventions: Other: Telehealth-based instructional visit and receive routine instructions

INTERVENTIONS:
Other: Receive routine instructions — Study subjects randomized to this arm will receive a mailed myLab Box kit with instructions on HPV self-collection and postage to be shipped directly to the commercial lab. It should take less than 5 minutes to collect the sample.
  Arms: Receive routine instructions
Other: Telehealth-based instructional visit and receive routine instructions — Study subjects randomized to this arm will similarly receive a mailed myLab Box kit and also undergo a brief 5-10" telehealth instructional visit via video conference.
  Arms: Telehealth Visit

SUMMARY:
This study aims to compare the efficacy and participant experience of telehealth-based, self-collected cervical cancer screening to mail-based, self-collected cervical cancer screening across the adult female screening lifespan. This will be done by evaluating sufficient Human papillomavirus (HPV) sample collection and determining preference for self-collection verses provider collection, comparing role of telehealth in pre- and post- menopausal women's comfort with self-collection, comparing self-collection completion rates for women with and without telehealth visits.

DETAILED DESCRIPTION:
This will be a prospective, randomized study of women ages 25 and older, stratified by menopausal status (defined as 12 months or greater without menses or time at which both ovaries have been surgically removed), who are eligible for cervical cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a cervix who are eligible for primary HPV testing (age 25 and older) according to national cervical cancer screening guidelines.
* Pregnant women are eligible for participation in this study as the collection process poses no threat to the woman or her fetus.

Exclusion Criteria:

* Individuals without a cervix
* Have had prior pelvic radiation therapy or brachytherapy
* Active or former diagnosis of ovarian, uterine, or cervical cancer unless determined eligible by PI upon further review of history and treatment
* Individuals less than age 25 or no longer eligible/recommended to undergo cervical cancer screening
* Adults who are unable to consent or are decisionally impaired
* Individuals who are not English speaking

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Proportion of participants preferring self-collection to provider collection | Post-intervention: 2 weeks after receipt of test results
  In follow-up survey, participants will indicate how the would prefer to have their next cervical cancer screening performed: by their healthcare provider or by self-testing.

SECONDARY OUTCOMES:
Median perceived difficulty understanding self-collection instructions | Post-intervention: 2 weeks after receipt of test results
  In follow-up survey, participants will indicate how difficult the self-collection instructions were to understand, on a 10-point Likert scale.
Median discomfort level with self-collection | Post-intervention: 2 weeks after receipt of test results
  In follow-up survey, participants will indicate how much discomfort their experienced during self-collection, on a 10-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Bruegl, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States